CLINICAL TRIAL: NCT05061134
Title: A Randomised, Open-Label, Phase 2 Study of Ceralasertib Monotherapy and Ceralasertib Plus Durvalumab in Patients With Unresectable or Advanced Melanoma and Primary or Secondary Resistance to PD-(L)1 Inhibition
Brief Title: A Study of Ceralasertib Monotherapy and Ceralasertib Plus Durvalumab in Patients With Melanoma and Resistance to PD-(L)1 Inhibition
Acronym: MONETTE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D533AC00001; 2024-512378-91-00 (Registry Identifier: CTIS); 2021-001722-21 (EudraCT Number)
Record Dates: First submitted 2021-09-22; First posted 2021-09-29 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Melanoma
Keywords: Unresectable or Advanced Melanoma; Efficacy; Safety
MeSH Terms: conditions — Melanoma | interventions — ceralasertib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Main study: Ceralasertib + Durvalumab (Experimental): Participants will receive ceralasertib on Days 1 to 7 plus durvalumab Day 8, once in 28 days (Q28D), until progressive disease, unacceptable toxicity, withdrawal of consent, or if a study treatment discontinuation criterion is met.
  Interventions: Drug: Ceralasertib; Biological: Durvalumab
- Main study: Ceralasertib (Experimental): Participants will receive ceralasertib on Days 1 to 7, Q28D, until progressive disease, unacceptable toxicity, withdrawal of consent, or if a study treatment discontinuation criterion is met.
  Interventions: Drug: Ceralasertib
- Biopsy Sub-study: Ceralasertib + Durvalumab (Experimental): From Cycle 1, participants will receive combination of ceralasertib twice daily (BD) Days 1 to 7 plus durvalumab Day 8, Q28D, until progressive disease, unacceptable toxicity, withdrawal of consent, or a study treatment discontinuation criterion is met.
  Interventions: Drug: Ceralasertib; Biological: Durvalumab
- Biopsy study: Ceralasertib (Experimental): During Cycle 0, participants will receive ceralasertib on Days 1 to 7, followed by an off-treatment period between Days 8 to 28.
  Interventions: Drug: Ceralasertib

INTERVENTIONS:
Drug: Ceralasertib — Ceralasertib (240 mg) will be administered orally twice daily.
Biological: Durvalumab — Durvalumab (1500 mg) will be administered intravenously once every 28 days for participants who weight above > 30 kgs. For participants who weigh below ≤ 30 kgs, weight-based dosing equivalent to 20 mg/kg of durvalumab will be administered.
  Arms: Biopsy Sub-study: Ceralasertib + Durvalumab; Main study: Ceralasertib + Durvalumab

SUMMARY:
Main study: This is an open-label, phase 2 study that aims to evaluate the efficacy and safety/tolerability of ceralasertib, when administered as monotherapy and in combination with durvalumab in participants with unresectable or advanced melanoma and primary or secondary resistance to PD-(L)1 inhibition.

DETAILED DESCRIPTION:
Biopsy sub-study: This is an open-label, non-randomised, sub-study planned in participants suitable for 3 mandatory biopsies. Serial tumour biopsies are mandated in participants recruited into the sub-study and will be taken at baseline during the screening period, during treatment with ceralasertib monotherapy and during the off-treatment period of ceralasertib monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically or cytologically confirmed diagnosis of unresectable or metastatic melanoma of cutaneous, acral or mucosal subtype
* Availability of an archival tumour sample and a fresh tumour biopsy taken at screening
* Patient must have received at least 1 prior immunotherapy (anti-PD-(L)1 ± anti-CTLA-4 [Cytotoxic T-lymphocyte-associated protein 4]) for a minimum of 6 weeks and no more than 2 prior regimens in the metastatic setting. Patients must have confirmed progression during treatment with a PD-(L)1 inhibitor +/- a CTLA-4 inhibitor.
* The interval between the last dose of anti-PD-(L)1, BRAF/MEK (B-Rapidly Accelerated Fibrosarcoma gene/mitogen-activated protein kinase gene) inhibitor and the first dose of the study regimen must be a minimum of 14 days
* Measurable disease by RECIST 1.1.
* Patients must have a life expectancy ≥3 months from proposed first dose date.
* Biopsy Sub-study: Consent to the provision of 3 mandatory tumour biopsies.

Exclusion Criteria:

* Patients must not have experienced a toxicity that led to permanent discontinuation of prior checkpoint inhibitors (CPI) treatment.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 3 years before the first dose of study treatment
* Uveal melanoma
* Must not have experienced a Grade ≥ 3 immune-related AE or an immune-related neurologic or ocular AE of any grade while receiving prior immunotherapy
* History of symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Patients with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be permitted upon discussion with the study clinical lead.
* History of organ transplant that requires use of immunosuppressive medications
* Inadequate bone marrow and impaired hepatic or renal function
* Known active infection requiring systemic therapy, active hepatitis infection, positive hepatitis C virus antibody, hepatitis B virus (HBV) surface antigen or HBV core antibody (anti-HBc), at screening
* Patients with confirmed COVID-19 infection by polymearse chain reaction test who have not made a full recovery.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2026-11-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (6):
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, Tampa, Florida
  - Research Site, Lutherville-Timonium, Maryland
  - Research Site, Nashville, Tennessee
- Australia (4):
  - Research Site, Darlinghurst
  - Research Site, East Melbourne
  - Research Site, Herston
  - Research Site, Woolloongabba
- Belgium (4):
  - Research Site, Belgium
  - Research Site, Bruges
  - Research Site, Ghent
  - Research Site, Leuven
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Ste-Foy, Quebec
- France (9):
  - Research Site, Bobigny
  - Research Site, Boulogne-Billancourt
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Germany (10):
  - Research Site, Berlin
  - Research Site, Buxtehude
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Kiel
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Regensburg
  - Research Site, Schwerin
  - Research Site, Tübingen
- Italy (7):
  - Research Site, Candiolo
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Perugia
  - Research Site, Roma
  - Research Site, Siena
- Poland (6):
  - Research Site, Brzozów
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
- South Korea (2):
  - Research Site, Goyang
  - Research Site, Seoul
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Pozuelo de Alarcón
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Chelsea
  - Research Site, Manchester
  - Research Site, Northwood

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D533AC00001_CSP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D533AC00001&attachmentIdentifier=09aadb67-9bca-4814-8a11-14413dcec89d&fileName=D533AC00001_CSP_Redacted.pdf&versionIdentifier=
- See also: D533AC00001_SAP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D533AC00001&attachmentIdentifier=8d2cd097-59f9-4306-beb0-6c9c8384bddb&fileName=D533AC00001_SAP_Redacted.pdf&versionIdentifier=
- See also: D533AC00001_CSR synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D533AC00001&attachmentIdentifier=ade8f993-e385-4f2c-bdfb-6bc468c0cff9&fileName=D533AC00001_CSR_synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 11 Aug 2022 (first participants enrolled) to 12 Apr 2024 (primary completion date). The study was conducted in 11 countries.
Pre-assignment Details: Participants who met the inclusion criteria and none of the exclusion criteria were enrolled to the study. Informed consent forms (ICFs) was signed prior to screening procedures. All study assessments were performed as per the Schedule of Activities.
Groups:
- Main Study: Ceralasertib + Durvalumab: Participants received ceralasertib 240 milligrams (mg) orally twice daily (BD) for 7 consecutive days (Days 1 to 7), and on Day 8, participants received 1500 mg durvalumab as an intravenous (IV) infusion once in every 28 days. This 28-day cycle was repeated until progressive disease, unacceptable toxicity, withdrawal of consent, or if a study treatment discontinuation criterion was met.
- Main Study: Ceralasertib Monotherapy: Participants received ceralasertib monotherapy 240 mg orally BD from Days 1 to 7, once in every 28 days. This 28-day cycle was repeated until progressive disease, unacceptable toxicity, withdrawal of consent, or if a study treatment discontinuation criterion was met.
- Biopsy Study: Ceralasertib + Durvalumab: Participants received ceralasertib monotherapy 240 mg orally BD for 7 consecutive days (Days 1 to 7) on Cycle 0.
  Onwards Cycle 1, participants received ceralasertib 240 mg orally BD for 7 consecutive days (Days 1 to 7) plus durvalumab 1500 mg as IV infusion on Day 8 once in every 28 days. This 28-day cycle was repeated until progressive disease, unacceptable toxicity, withdrawal of consent, or if a study treatment discontinuation criterion was met.
Period: Overall Study
Arm/Group | Main Study: Ceralasertib + Durvalumab | Main Study: Ceralasertib Monotherapy | Biopsy Study: Ceralasertib + Durvalumab
Started | 100 | 51 | 43
Completed | 0 | 0 | 0
Not Completed | 100 | 51 | 43
Not completed — Patients ongoing in the study at data cut-off (DCO) of 12-April-2024 | 19 | 3 | 6
Not completed — Subject not treated | 0 | 0 | 2
Not completed — Other | 0 | 0 | 9
Not completed — Withdrawal by Subject | 9 | 8 | 5
Not completed — Study Terminated by Sponsor | 22 | 14 | 7
Not completed — Progressive Disease | 1 | 2 | 0
Not completed — Patient Is on Survival Follow Up Beyond DCO | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Disease progression | 1 | 0 | 0
Not completed — Death | 43 | 23 | 14
Not completed — Database lock | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For main study: Full analysis set (FAS) included all participants who were randomized in the study.
  For biopsy study: Safety analysis set included all participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study: Ceralasertib + Durvalumab | Main Study: Ceralasertib Monotherapy | Biopsy Study: Ceralasertib + Durvalumab | Total
Number analyzed (Participants) | 100 | 51 | 41 | 192
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (13.6) | 62.9 (12.6) | 61.4 (11.9) | 62.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 22 | 16 | 80
  Male | 58 | 29 | 25 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 79 | 39 | 31 | 149
  Asian | 9 | 7 | 0 | 16
  Other | 2 | 1 | 0 | 3
  Not reported | 10 | 4 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants who had a complete response (CR) or partial response (PR) prior to any evidence of progression (as defined by Response Evaluation Criteria in Solid Tumours [RECIST] 1.1) that is confirmed at least 4 weeks later.
  As per planned in protocol, this outcome measure was assessed only for main study.
Time Frame: Cycle 1 Day 1 (Each Cycle is 28 days) until objective disease progression or the last evaluable assessment in the absence of progression, or data cut-off (1 year 8 months)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Participants were summarized according to the actual treatment received.
  Here, two participants, who were randomized to the Main Study: Ceralasertib + Durvalumab group, started with ceralasertib but did not receive durvalumab. Hence, they are summarized in the Main Study: Ceralasertib monotherapy group (actual treatment group) for the outputs presented in the safety analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Main Study: Ceralasertib + Durvalumab | Main Study: Ceralasertib Monotherapy
Number analyzed (Participants) | 97 | 52
Percentage of participants | 9.3 [4.3 to 16.9] | 5.8 [1.2 to 15.9]

2. Primary Outcome: Biopsy Study: Change From Baseline in CD8+ T-cells Tumour Infiltration-area in the Center Tumor Region
Description: Changes in CD8+ T-cell infiltration of tumours induced by ceralasertib monotherapy was assessed in baseline, on-treatment and off-treatment tumour biopsies As per planned in protocol, this outcome measure was assessed only for biopsy study.
Time Frame: Baseline, On-treatment (Cycle 0 Day 7), and Off-treatment (Cycle 0 Day 15-28) (each cycle is 28 days)
Population: Pharmacodynamic (PD) analysis set included all participants who received at least 1 dose of study treatment with at least 1 reportable post-baseline pharmacodynamic measurement. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 23
Percent change
  On-treatment: number analyzed (Participants) | 18
  On-treatment | -0.976 (2.920)
  Off-treatment | -0.451 (1.357)

3. Secondary Outcome: Main Study and Biopsy Study: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documented confirmed response until date of documented progression per RECIST 1.1 or death due to any cause.
  For main study BICR data is presented, and for Biopsy sub study, investigator assessment data has been presented.
Time Frame: Cycle 1 Day 1 (each cycle is 28 days) until date of documented progression or data cut-off (2 years), whichever occurred first
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Participants were summarized according to the actual treatment received. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure and participants with objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: Ceralasertib + Durvalumab | Main Study: Ceralasertib Monotherapy | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 9 | 3 | 2
Months | NA [7.5 to NA] — Here, NA indicate that median and upper limit of 95% CI were not evaluable due to insufficient number of participants with events. | NA [5.6 to NA] — Here, NA indicate that median and upper limit of 95% CI were not evaluable due to insufficient number of participants with events. | NA [5.8 to NA] — Here, NA indicate that median and upper limit of 95% CI were not evaluable due to insufficient number of participants with events.

4. Secondary Outcome: Main Study and Biopsy Study: Time to Response
Description: Time to response was defined as the time from randomization until the date of first documented objective response, which is subsequently confirmed per RECIST 1.1.
  For main study blinded independent central review (BICR) data is presented, and for Biopsy sub study, investigator assessment data has been presented.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: Ceralasertib + Durvalumab | Main Study: Ceralasertib Monotherapy | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 9 | 3 | 2
Months | 3.5 [1.7 to 5.6] | 3.6 [2.4 to NA] — Here, NA indicate that upper limit of 95% CI was not evaluable due to insufficient number of participants with events. | 3.7 [2.7 to NA] — Here, NA indicate that upper limit of 95% CI was not evaluable due to insufficient number of participants with events.

5. Secondary Outcome: Main Study and Biopsy Study: Percentage Change From Baseline in Tumour Size
Description: Percentage change from baseline in target lesion (TL) tumour size was assessed. Tumour size is the sum of the longest diameters of the target lesions. The percentage change from baseline in TL tumour size at post-baseline assessment is obtained for each participants taking the difference between the sum of the TLs at post baseline assessment and the sum of the TLs at baseline divided by the sum of the TLs at baseline times 100. Percentage change from baseline at 16 weeks for main study and 20 weeks for biopsy study in sum of target lesions has been presented.
  For main study, BICR data is presented, and for Biopsy sub study, investigator assessment data has been presented.
Time Frame: Main Study: at 16 weeks; Biopsy study: at 20 weeks
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Participants were summarized according to the actual treatment received. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Main Study: Ceralasertib + Durvalumab | Main Study: Ceralasertib Monotherapy | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 76 | 41 | 29
Percentage change from baseline | 15.80 (38.14) | 11.25 (33.99) | 17.93 (38.46)

6. Secondary Outcome: Main Study and Biopsy Study: Progression Free Survival (PFS)
Description: PFS was defined as time from randomization until progression per RECIST 1.1 or death due to any cause.
  For main study BICR data is presented, and for Biopsy sub study, investigator assessment data has been presented.
Time Frame: as for outcome 3
Population: For main study: Full analysis set included all participants who were randomized in the study.
  For biopsy study: Safety analysis set included all participants who received at least 1 dose of study treatment. Participants were summarized according to the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: Ceralasertib + Durvalumab | Main Study: Ceralasertib Monotherapy | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 100 | 51 | 41
Months | 2.00 [1.91 to 3.52] | 1.94 [1.91 to 3.06] | 2.83 [2.76 to 4.47]

7. Secondary Outcome: Main Study and Biopsy Study: Overall Survival (OS)
Description: OS was defined as time from date of randomization until the date of death due to any cause.
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Main Study: Ceralasertib + Durvalumab | Main Study: Ceralasertib Monotherapy | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 100 | 51 | 41
Months | 16.00 [10.48 to NA] — Here, NA indicate that upper limit of 95% CI was not evaluable due to insufficient number of participants with events and due to the duration of follow-up. | 12.32 [9.46 to NA] — Here, NA indicate that upper limit of 95% CI was not evaluable due to insufficient number of participants with events and due to the duration of follow-up. | NA [10.18 to NA] — Here, NA indicate that median and upper limit of 95% CI was not evaluable due to insufficient number of participants with events and due to the duration of follow-up.

8. Secondary Outcome: Main Study: Plasma Concentration of Ceralasertib
Description: Pharmacokinetic (PK) of ceralasertib alone and when in combination with durvalumab was assessed.
Time Frame: From Cycle 1 to Cycle 4: Day 7 and Day 8 of each cycle (each cycle is 28 days); 90 days follow-up
Population: The PK analysis set included all dosed participants with reportable ceralasertib or durvalumab plasma concentrations. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure and 'number analyzed in each row' signifies the participants with available data that were analyzed for specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Main Study: Ceralasertib + Durvalumab | Main Study: Ceralasertib Monotherapy
Number analyzed (Participants) | 85 | 41
Nanograms per milliliter (ng/mL)
  Cycle 1 Day 7: pre-dose: number analyzed (Participants) | 79 | 39
  Cycle 1 Day 7: pre-dose | 4621 (68.34) | 4789 (52.03)
  Cycle 1 Day 7: 1 hour post-dose | 8304 (44.69) | 8010 (53.84)
  Cycle 1 Day 8: pre-dose: number analyzed (Participants) | 3 | 0
  Cycle 1 Day 8: pre-dose | 78.10 (43.66) |
  Cycle 1 Day 8: 1 hour post-dose: number analyzed (Participants) | 82 | 0
  Cycle 1 Day 8: 1 hour post-dose | 379600 (23.05) |
  Cycle 2 Day 7: pre-dose: number analyzed (Participants) | 73 | 36
  Cycle 2 Day 7: pre-dose | 4487 (70.46) | 4101 (40.53)
  Cycle 2 Day 7: 1 hour post-dose: number analyzed (Participants) | 82 | 32
  Cycle 2 Day 7: 1 hour post-dose | 7735 (53.09) | 7984 (45.39)
  Cycle 2 Day 8: pre-dose: number analyzed (Participants) | 63 | 0
  Cycle 2 Day 8: pre-dose | 67170 (47.38) |
  Cycle 2 Day 8: 1 hour post-dose: number analyzed (Participants) | 73 | 0
  Cycle 2 Day 8: 1 hour post-dose | 425900 (36.73) |
  Cycle 3 Day 7: pre-dose: number analyzed (Participants) | 47 | 21
  Cycle 3 Day 7: pre-dose | 4269 (44.72) | 4045 (51.17)
  Cycle 3 Day 7: 1 hour post-dose: number analyzed (Participants) | 50 | 25
  Cycle 3 Day 7: 1 hour post-dose | 7072 (41.81) | 7799 (41.76)
  Cycle 3 Day 8: pre-dose: number analyzed (Participants) | 45 | 0
  Cycle 3 Day 8: pre-dose | 105100 (50.26) |
  Cycle 3 Day 8: 1 hour post-dose: number analyzed (Participants) | 50 | 0
  Cycle 3 Day 8: 1 hour post-dose | 460800 (26.48) |
  Cycle 4 Day 7: pre-dose: number analyzed (Participants) | 0 | 1
  Cycle 4 Day 7: pre-dose |  | NA (NA) — Here, geometric mean and geometric Coefficient of Variation could not be calculated due to insufficient number of participants as pre-specified in the SAP.
  Cycle 4 Day 7: 1 hour post-dose: number analyzed (Participants) | 0 | 3
  Cycle 4 Day 7: 1 hour post-dose |  | 7273 (33.82)
  90 Days Follow-up: number analyzed (Participants) | 8 | 0
  90 Days Follow-up | 23830 (79.06) |

9. Secondary Outcome: Main Study and Biopsy Study: Number of Participants With Adverse Events (AEs)
Description: The safety and tolerability of ceralasertib monotherapy and ceralasertib plus durvalumab in participants with unresectable or advanced melanoma and primary or secondary resistance to a programmed death ligand 1 (PD-[L] 1) inhibitor was assessed.
  The grading scales found in the revised National Cancer Institute CTCAE latest version was utilized for all events with an assigned CTCAE grading. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 where Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL; Grade 4: Life-threatening, urgent intervention required; Grade 5: Death related to AE.
Time Frame: From screening (Day -28 to -1) until Safety follow-up (30 days after last dose of Ceralasertib monotherapy or 90 days after last dose of Ceralasertib+Durvalumab combination) or data cut-off (2 years), whichever occurred first
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Ceralasertib + Durvalumab | Main Study: Ceralasertib Monotherapy | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 97 | 52 | 41
Participants
  Any AE | 92 | 45 | 39
  Any AE possibly related to treatment | 74 | 36 | 29
  Any AE of >= CTCAE grade 3 | 34 | 16 | 13
  Any AE of >= CTCAE grade 3, possibly related to treatment | 17 | 9 | 4
  Any SAE | 19 | 5 | 9
  Any SAE possibly related to treatment | 3 | 2 | 0
  Any SAE of >= CTCAE grade 3 | 16 | 3 | 9
  Any SAE of >= CTCAE grade 3, possibly related to treatment | 3 | 0 | 0
  Any SAE with outcome death | 0 | 0 | 1
  Any SAE with outcome death, possibly related to treatment | 0 | 0 | 0
  Any AE leading to discontinuation of treatment | 1 | 1 | 1
  Any AE leading to discontinuation of treatment, possibly related to treatment | 1 | 1 | 1
  Any AE leading to drug interruption of treatment | 8 | 3 | 8
  Any AE leading to dose reduction of treatment | 10 | 6 | 3
  Any AE leading to dose modification of treatment | 14 | 8 | 9
  Any SAE leading to discontinuation of treatment | 0 | 0 | 0
  Any SAE leading to discontinuation of treatment, possibly related to treatment | 0 | 0 | 0
  Any SAE leading to drug interruption of treatment | 5 | 1 | 4
  Any SAE leading to dose reduction of treatment | 2 | 0 | 0
  Any SAE leading to dose modification of treatment | 5 | 1 | 4
  Any AE of >= CTCAE grade 3, possibly related to Ceralasertib | 16 | 9 | 4
  Any AE of >= CTCAE grade 3, possibly related to Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any AE of >= CTCAE grade 3, possibly related to Durvalumab | 5 |  | 1
  Any SAE possibly related to Ceralasertib | 3 | 2 | 0
  Any SAE possibly related to Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any SAE possibly related to Durvalumab | 1 |  | 0
  Any SAE of >= CTCAE grade 3, possibly related to Ceralasertib | 3 | 0 | 0
  Any SAE of >= CTCAE grade 3, possibly related to Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any SAE of >= CTCAE grade 3, possibly related to Durvalumab | 1 |  | 0
  Any SAE with outcome death, possibly related to Ceralasertib | 0 | 0 | 0
  Any SAE with outcome death, possibly related to Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any SAE with outcome death, possibly related to Durvalumab | 0 |  | 0
  Any AE leading to discontinuation of Ceralasertib | 1 | 1 | 1
  Any AE leading to discontinuation of Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any AE leading to discontinuation of Durvalumab | 0 |  | 1
  Any AE leading to discontinuation of Ceralasertib, possibly related to Ceralasertib | 1 | 1 | 1
  Any AE leading to discontinuation of Durvalumab, possibly related to Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any AE leading to discontinuation of Durvalumab, possibly related to Durvalumab | 0 |  | 1
  Any AE leading to drug interruption of Ceralasertib | 6 | 3 | 8
  Any AE leading to drug interruption of Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any AE leading to drug interruption of Durvalumab | 5 |  | 2
  Any AE leading to dose reduction of Ceralasertib | 10 | 6 | 3
  Any AE leading to dose reduction of Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any AE leading to dose reduction of Durvalumab | 0 |  | 0
  Any AE leading to dose modification of Ceralasertib | 13 | 8 | 9
  Any AE leading to dose modification of Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any AE leading to dose modification of Durvalumab | 5 |  | 2
  Any SAE leading to discontinuation of Ceralasertib | 0 | 0 | 0
  Any SAE leading to discontinuation of Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any SAE leading to discontinuation of Durvalumab | 0 |  | 0
  Any SAE leading to discontinuation of Ceralasertib, possibly related to Ceralasertib | 0 | 0 | 0
  Any SAE leading to discontinuation of Durvalumab, possibly related to Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any SAE leading to discontinuation of Durvalumab, possibly related to Durvalumab | 0 |  | 0
  Any SAE leading to drug interruption of Ceralasertib | 4 | 1 | 4
  Any SAE leading to drug interruption of Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any SAE leading to drug interruption of Durvalumab | 3 |  | 1
  Any SAE leading to dose reduction of Ceralasertib | 2 | 0 | 0
  Any SAE leading to dose reduction of Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any SAE leading to dose reduction of Durvalumab | 0 |  | 0
  Any SAE leading to dose modification of Ceralasertib | 4 | 1 | 4
  Any SAE leading to dose modification of Durvalumab: number analyzed (Participants) | 97 | 0 | 41
  Any SAE leading to dose modification of Durvalumab | 3 |  | 1

10. Secondary Outcome: Biopsy Study: Number of Participants With Presence of PD-L1 Overtime
Description: Pre-treatment presence and/or on-treatment and/or off-treatment changes in PD-L1 was assessed to collect tumour tissue samples, or utilise residual samples, for the analysis of tumoural biomarkers that change following treatment with ceralasertib was assessed.
  As per planned in protocol, this outcome measure was assessed only for biopsy study. The number of patients with PD-L1 expression <1% and >= 1% has been presented.
Time Frame: Baseline, On-treatment (Cycle 0 Day 7); Off-treatment (Cycle 0 Day 15-28) (each cycle is 28 days)
Population: The PD analysis set included all participants who received at least 1 dose of study treatment with at least 1 reportable post-baseline pharmacodynamic measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 36
Participants
  Tumor Positive Membrane score: Baseline: <1% PD-L1 expression | 22
  Tumor Positive Membrane score: Baseline: >=1% PD-L1 expression | 8
  Tumor Positive Membrane score: On-treatment (Cycle 0 Day 7): <1% PD-L1 expression | 14
  Tumor Positive Membrane score: On-treatment (Cycle 0 Day 7): >=1% PD-L1 expression | 6
  Tumor Positive Membrane score: Off-treatment (Cycle 0 Day 15-28): <1% PD-L1 expression | 17
  Tumor Positive Membrane score: Off-treatment (Cycle 0 Day 15-28): >=1% PD-L1 expression | 8
  Tumor Positive Membrane score: Off-treatment (Cycle 0 Day 15-28): unknown | 1
  Tumor Area Positivity score: Baseline:<1% PD-L1 expression | 12
  Tumor Area Positivity score: Baseline: >=1% PD-L1 expression | 18
  Tumor Area Positivity score: On-treatment (Cycle 0 Day 7): <1% PD-L1 expression | 10
  Tumor Area Positivity score: On-treatment (Cycle 0 Day 7): >=1% PD-L1 expression | 10
  Tumor Area Positivity score: Off-treatment (Cycle 0 Day 15-28): <1% PD-L1 expression | 9
  Tumor Area Positivity score: Off-treatment (Cycle 0 Day 15-28): >=1% PD-L1 expression | 16
  Tumor Area Positivity score: Off-treatment (Cycle 0 Day 15-28): unknown | 1

11. Secondary Outcome: Biopsy Study: Number of Participants With Presence of pRAD50
Description: Pre-treatment presence and/or on-treatment and/or off-treatment changes in pRAD50 was assessed to collect tumour tissue samples, or utilise residual samples, for the analysis of tumoural biomarkers that change following treatment with ceralasertib was assessed.
  As per planned in protocol, this outcome measure was assessed only for biopsy study.
Time Frame: On-treatment (Cycle 0 Day 7); Off-treatment (Cycle 0 Day 15-28) (each cycle is 28 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 36
Participants
  Baseline | 29
  On-treatment (Cycle 0 Day 7) | 18
  Off-treatment (Cycle 0 Day 15-28) | 25

12. Secondary Outcome: Biopsy Study: Change From Baseline in Proliferation (Using Ki67+ Marker) of Carcinoma and/or Immune Cells (Including CD8+ T Cells) - Cell Density in Center Tumour Region
Description: Changes in the proliferation of carcinoma and/or immune cells within tumours induced by ceralasertib monotherapy was assessed.
  As per planned in protocol, this outcome measure was assessed only for biopsy study.
Time Frame: Baseline, On-treatment (Cycle 0 Day 7); Off-treatment (Cycle 0 Day 15-28) (each cycle is 28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Change in cells per mm2
Arm/Group | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 23
Change in cells per mm2
  CD8+ IHC: On-treatment (Cycle 0 Day 7): number analyzed (Participants) | 18
  CD8+ IHC: On-treatment (Cycle 0 Day 7) | -183.589 (740.398)
  CD8+ IHC: Off-treatment (Cycle 0 Day 15-28) | -85.259 (396.091)
  Ki67+ IHC: On-treatment (Cycle 0 Day 7): number analyzed (Participants) | 18
  Ki67+ IHC: On-treatment (Cycle 0 Day 7) | -355.399 (461.152)
  Ki67+ IHC: Off-treatment (Cycle 0 Day 15-28) | 47.656 (1041.627)

13. Primary Outcome: Biopsy Study: Change From Baseline in CD8+ T-cells Tumour Infiltration-area in the Invasive Margin Region
Description: Changes in CD8+ T-cell infiltration of tumours induced by ceralasertib monotherapy was assessed in baseline and off-treatment tumour biopsies As per planned in protocol, this outcome measure was assessed only for biopsy study.
Time Frame: Baseline, Off-treatment (Cycle 0 Day 15-28) (each cycle is 28 days)
Population: The PD analysis set included all participants who received at least 1 dose of study treatment with at least 1 reportable post-baseline pharmacodynamic measurement. Here, 'number of participants analyzed' specifies all participants who were evaluated for this outcome measure.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 1
Percent change | NA [-0.73 to -0.73] — As pre-specified in statistical analysis plan (SAP), median is not calculable due to insufficient number of participants.

14. Primary Outcome: Biopsy Study: Change From Baseline in CD8+ T-cells Tumour Infiltration-density in the Center Tumor Region
Description: as for outcome 2
Time Frame: Baseline, On-treatment (Cycle 0 Day 7), and Off-treatment (Cycle 0 Day 15-28) (each cycle is 28 days)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Change in cells per mm^2
Arm/Group | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 23
Change in cells per mm^2
  On-treatment: number analyzed (Participants) | 18
  On-treatment | -183.589 (740.398)
  Off-treatment | -85.259 (396.091)

15. Primary Outcome: Biopsy Study: Change From Baseline in CD8+ T-cells Tumour Infiltration-density in the Invasive Margin Region
Description: as for outcome 13
Time Frame: Baseline, and Off-treatment (Cycle 0 Day 15-28) (each cycle is 28 days)
Population: as for outcome 13
Measure: Median (Full Range); unit: Change in cells per mm^2
Arm/Group | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 1
Change in cells per mm^2 | NA [-235.53 to -235.53] — As pre-specified in statistical analysis plan (SAP), median is not calculable due to insufficient number of participants.

16. Secondary Outcome: Biopsy Study: Change From Baseline in Proliferation (Using Ki67+ Marker) of Carcinoma and/or Immune Cells (Including CD8+ T Cells) - Cell Density in Invasive Margin Region
Description: as for outcome 12
Time Frame: Baseline, On-treatment (Cycle 0 Day 7); Off-treatment (Cycle 0 Day 15-28) (each cycle is 28 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: Change in cells per mm2
Arm/Group | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 1
Change in cells per mm2
  CD8+ IHC: Off-treatment (Cycle 0 Day 15-28) | NA [-235.53 to -235.53] — As pre-specified in SAP, median is not calculable due to insufficient number of participants.
  Ki67+ IHC: Off-treatment (Cycle 0 Day 15-28) | NA [194.39 to 194.39] — As pre-specified in SAP, median is not calculable due to insufficient number of participants.

17. Secondary Outcome: Biopsy Study: Change From Baseline in Proliferation (Using Ki67+ Marker) of Carcinoma and/or Immune Cells (Including CD8+ T Cells) - Area in Centre Tumour Region
Description: as for outcome 12
Time Frame: Baseline, On-treatment (Cycle 0 Day 7); Off-treatment (Cycle 0 Day 15-28) (each cycle is 28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 23
Percent change
  CD8+ cells: On-treatment (Cycle 0 Day 7): number analyzed (Participants) | 18
  CD8+ cells: On-treatment (Cycle 0 Day 7) | -0.976 (2.920)
  CD8+ cells: Off-treatment (Cycle 0 Day 15-28) | -0.451 (1.357)
  Ki67+ Cells: On-treatment (Cycle 0 Day 7): number analyzed (Participants) | 18
  Ki67+ Cells: On-treatment (Cycle 0 Day 7) | -1.953 (2.616)
  Ki67+ Cells: Off-treatment (Cycle 0 Day 15-28) | 0.754 (6.931)

18. Secondary Outcome: Biopsy Study: Change From Baseline in Proliferation (Using Ki67+ Marker) of Carcinoma and/or Immune Cells (Including CD8+ T Cells) - Area in Invasive Margin Region
Description: as for outcome 12
Time Frame: Baseline, On-treatment (Cycle 0 Day 7); Off-treatment (Cycle 0 Day 15-28) (each cycle is 28 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: Percent change
Arm/Group | Biopsy Study: Ceralasertib + Durvalumab
Number analyzed (Participants) | 1
Percent change
  CD8+ cells: Off-treatment (Cycle 0 Day 15-28) | NA [-0.73 to -0.73] — As pre-specified in SAP, median is not calculable due to insufficient number of participants.
  Ki67+ Cells: Off-treatment (Cycle 0 Day 15-28) | NA [1.08 to 1.08] — As pre-specified in SAP, median is not calculable due to insufficient number of participants.

ADVERSE EVENTS:
Time Frame: From screening (Day -28 to -1) until Safety follow-up (30 days after last dose of Ceralasertib monotherapy or 90 days after last dose of Ceralasertib+Durvalumab combination) or data cut-off (2 years), whichever occurred first
Description: Safety analysis set included all participants who received at least 1 dose of study treatment. Participants were summarized according to the actual treatment received.
  All-cause mortality for main study was assessed in full analysis set (FAS). The FAS included all participants who were randomized in the study.
Arm/Group | Main Study: Ceralasertib + Durvalumab | Main Study: Ceralasertib Monotherapy | Biopsy Study: Ceralasertib + Durvalumab
All-Cause Mortality (participants affected / at risk) | 43/100 | 23/51 | 14/41
Serious Adverse Events (participants affected / at risk) | 19/97 | 5/52 | 9/41
Other Adverse Events (participants affected / at risk) | 86/97 | 43/52 | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Ceralasertib + Durvalumab (N=97) | Main Study: Ceralasertib Monotherapy (N=52) | Biopsy Study: Ceralasertib + Durvalumab (N=41)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Proteus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Ceralasertib + Durvalumab (N=97) | Main Study: Ceralasertib Monotherapy (N=52) | Biopsy Study: Ceralasertib + Durvalumab (N=41)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (12) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 35 (55) | 9 (12) | 15 (20)
Leukopenia (Blood and lymphatic system disorders) | 5 (8) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 7 (17) | 2 (3) | 4 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (14) | 3 (6) | 5 (13)
Hypothyroidism (Endocrine disorders) | 1 (1) | 3 (6) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 20 (30) | 12 (14) | 11 (14)
Headache (Nervous system disorders) | 13 (29) | 3 (5) | 6 (7)
Hypertension (Vascular disorders) | 4 (5) | 4 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (10) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 10 (14) | 1 (2) | 6 (6)
Constipation (Gastrointestinal disorders) | 10 (11) | 1 (1) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 11 (19) | 6 (8) | 11 (15)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 1 (1) | 3 (6)
Nausea (Gastrointestinal disorders) | 50 (100) | 19 (25) | 20 (38)
Vomiting (Gastrointestinal disorders) | 21 (33) | 8 (9) | 13 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (23) | 5 (7) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 9 (12) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (8) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (15) | 5 (6) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 2 (2) | 4 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2) | 3 (4)
Asthenia (General disorders) | 22 (33) | 11 (13) | 8 (12)
Chills (General disorders) | 5 (8) | 0 (0) | 0 (0)
Fatigue (General disorders) | 19 (22) | 14 (17) | 10 (14)
Influenza like illness (General disorders) | 5 (6) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 11 (14) | 3 (3) | 3 (4)
Alanine aminotransferase increased (Investigations) | 7 (8) | 4 (4) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 8 (9) | 3 (3) | 4 (5)
C-reactive protein increased (Investigations) | 5 (8) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 10 (11) | 3 (3) | 7 (8)
Neutrophil count decreased (Investigations) | 2 (2) | 4 (6) | 0 (0)
Platelet count decreased (Investigations) | 10 (14) | 3 (4) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 4 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB.

DOCUMENTS (2):
  • Study Protocol (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT05061134/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT05061134/SAP_001.pdf